CLINICAL TRIAL: NCT00464659
Title: Comparison of the Evolution of Memory Deficit in Patients With Sleep Apnea Obstructive Syndrome (SAOS) Before and After "Effective" Versus Sham Treatment by Positive Pression Continues (PPC)
Brief Title: Protocol Memory Deficit in Patients With Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0629
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Memory Deficit
Keywords: Sleep apnea obstructive syndrome (SAOS); memory deficit; Continuous Positive Airway Pression (CPAP); Sham CPAP
MeSH Terms: conditions — Memory Disorders; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Effective CPAP treatment (Experimental): Effective Continuous Positive Airway Pressure treatment (CPAP) applied for 6 weeks
  Interventions: Device: Effective CPAP
- Sham CPAP treatment (Sham Comparator): Ineffective Continuous Positive Airway Pressure treatment (sham CPAP) applied for 6 weeks
  Interventions: Device: Sham CPAP

INTERVENTIONS:
Device: Effective CPAP — Auto-titrating CPAP machines (Remstar Auto; Philips Respironics, Murrysville, PA) provided by a home care company (Bastide Medical, France). Pressure was set between 6 and 14 cm of water
  Arms: Effective CPAP treatment
Device: Sham CPAP — Similar CPAP machine delivering a 4 cm of water pressure that was too low to suppress sleep respiratory events.
  Arms: Sham CPAP treatment

SUMMARY:
The main objective of this study is to evaluate the evolution of memory deficit (verbal episodic memory, procedural memory, working memory, short-term memory) in Sleep Apnea Obstructive Syndrome (SAOS) patients after treatment by Continuous Positive Airway Pressure treatment (CPAP). For thus, we will compare memory tests in two separate groups of SAOS patients with "effective " versus "ineffective" ( or sham) CPAP, before and 6 weeks after the beginning of the treatment. Thus we will assess the evolution of memory deficit, the effectiveness of the treatment on the evolution of memory deficit before and 6 weeks after the beginning of the treatment by "effective " versus "ineffective" CPAP.

We feel the results of the tests of memory will show greater memory disorders in patients with SAOS before beginning the treatment rather than six weeks afterwards. Thus we hypothesise that, after the treatment by "effective" CPAP, the patients with SAOS will have greater improvement of their memory disorders than those treated by "sham CPAP".

DETAILED DESCRIPTION:
We want to assess the evolution, before and 6 weeks after the beginning of the treatment, of the significant differences of the performances of the various memory tests evaluating several forms of memory (episodic memory, working memory, short-term memory and procedural memory) according to the treatment for patients with SAOS (effective versus sham).

ELIGIBILITY:
Inclusion Criteria:

* Major patients,
* agreeing,
* diagnosed suffering from the SAOS,
* regulation by the specialist in a treatment by CPAP,
* patients do not begin the treatment
* affiliated to the social security,
* fluent in French.

Exclusion Criteria:

* Patients presenting severe depressive disorders (HADS score>19),
* intellectual deterioration (MMS< 28),
* a functional failure of the dominant arm upper limb inhibiting realization of graphic tasks,
* an associated oxygen treatment,
* suffering from cancer,
* cerebro-vascular accident,
* pregnant or nursing women,
* adult under supervision or trusteeship,
* patients already included in another research protocol or in period of exclusion,
* antidepressant and anxiolytic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis JP Pépin, ProfessorPhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Laboratoire EFCR-Functional Cardio-Respiratory Exploration Laboratory, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data are anonymized

REFERENCES:
- [Background] Beebe DW, Gozal D. Obstructive sleep apnea and the prefrontal cortex: towards a comprehensive model linking nocturnal upper airway obstruction to daytime cognitive and behavioral deficits. J Sleep Res. 2002 Mar;11(1):1-16. doi: 10.1046/j.1365-2869.2002.00289.x. PMID 11869421
- [Background] Engleman HM, Douglas NJ. Sleep. 4: Sleepiness, cognitive function, and quality of life in obstructive sleep apnoea/hypopnoea syndrome. Thorax. 2004 Jul;59(7):618-22. doi: 10.1136/thx.2003.015867. PMID 15223874
- [Background] Farre R, Hernandez L, Montserrat JM, Rotger M, Ballester E, Navajas D. Sham continuous positive airway pressure for placebo-controlled studies in sleep apnoea. Lancet. 1999 Apr 3;353(9159):1154. doi: 10.1016/S0140-6736(99)01056-9. No abstract available. PMID 10209985
- [Background] Naegele B, Launois SH, Mazza S, Feuerstein C, Pepin JL, Levy P. Which memory processes are affected in patients with obstructive sleep apnea? An evaluation of 3 types of memory. Sleep. 2006 Apr;29(4):533-44. doi: 10.1093/sleep/29.4.533. PMID 16676787
- [Derived] Joyeux-Faure M, Naegele B, Pepin JL, Tamisier R, Levy P, Launois SH. Continuous positive airway pressure treatment impact on memory processes in obstructive sleep apnea patients: a randomized sham-controlled trial. Sleep Med. 2016 Aug;24:44-50. doi: 10.1016/j.sleep.2016.06.023. Epub 2016 Aug 23. PMID 27810185
- [Derived] Jullian-Desayes I, Tamisier R, Zarski JP, Aron-Wisnewsky J, Launois-Rollinat SH, Trocme C, Levy P, Joyeux-Faure M, Pepin JL. Impact of effective versus sham continuous positive airway pressure on liver injury in obstructive sleep apnoea: Data from randomized trials. Respirology. 2016 Feb;21(2):378-85. doi: 10.1111/resp.12672. Epub 2015 Nov 16. PMID 26567858